CLINICAL TRIAL: NCT05519501
Title: Randomized Controlled Clinical Investigation Evaluating the Effect of Adipose Tissue Processed With the SyntrFuge™ System in the Healing of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syntr Health Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHT-SYN-01
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Microsized Fat Tissue; Adipose Tissue; DFU; Wound Management
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SyntrFuge System (Experimental): Adipose tissue microsized via the SyntrFuge System
  Interventions: Device: SyntrFuge System
- Standard of Care (Other): Offloading
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: SyntrFuge System — Microsized Adipose Tissue
  Arms: SyntrFuge System
Procedure: Standard of Care — Offloading
  Arms: Standard of Care

SUMMARY:
This is a randomized controlled multi center study on diabetic patients with the aim of evaluating the efficacy of the adipose tissue processed with the SyntrFuge™ system in diabetic patients with diabetic foot ulcers. In particular, it will be evaluated whether the microsized fat graft will be able to shorten the healing times of these wounds. Patients will be randomized to the treatment group with adipose tissue processed with the SyntrFuge™ system (injection of autologous microsized adipose tissue) or to the control group represented by the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have Diabetic Foot Ulcer located at the plantar or dorsal aspect of the foot or the heel with a surface area of 1.0cm2 - 25cm2
2. Index ulcer has been present for greater than four weeks
3. Diabetics included will be those with HbA1c ≤ 12%
4. Subjects aged 18 - 85, inclusive
5. The target ulcer has been offloaded for at least 14 days

Exclusion Criteria:

1. Subjects without decisional capacity
2. Subjects unable to give informed, written consent
3. Subjects with active infection (redness, swelling, pain, suppuration)
4. Subjects with active osteomyelitis to the index ulcer
5. Subjects with previous treatment with Negative Pressure Wound Therapy, growth factors, radiation, hyperbaric O2, or bioengineered tissue product within 30 days of Screening
6. Subjects with a previous diagnosis of HIV or Hep C
7. Subject is pregnant or breast feeding
8. Subjects receiving oncological treatments ongoing or previous (past 5 years) and/or neoplastic lesions
9. Subjects under corticosteroid therapy, unless taking dose of 5mg/dl or less
10. Subjects with any other condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with study wound deemed closed at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Roanoke, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No